CLINICAL TRIAL: NCT04694872
Title: The Effects of Telerehabilitation-based Exercise Trainings on Gait and Balance in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Principla Investigator, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Istanbul University Cerrahpasa
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Tele-rehabilitation; Exercise; LSVT BIG
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a) TELEREHABILITATION BASED LSVT BIG TREATMENT GROUP (Experimental): It is planned to recruit 16 patients with Parkinson's Disease in this group. Exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week, 60 minutes a day, 4 weeks protocol respectively.
  Interventions: Other: Telerehabilitation Based LSVT BIG Exercise Protocol
- b) TELEREHABILITATION BASED FUNCTIONAL BALANCE AND MOBILITY EXERCISES GROUP (Active Comparator): It is planned to recruit 16 patients with Parkinson's Disease in this group. These exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week and 60 minutes a day for 4 weeks.
  Interventions: Other: Telerehabilitation Based Functional Balance and Mobility Exercise

INTERVENTIONS:
Other: Telerehabilitation Based LSVT BIG Exercise Protocol — Lee Silverman Voice Treatment-LOUD therapy is a protocol involving intensive speech therapy, which was initiated at the Lee Silverman Parkinson Center between 1987-1989 to heal hypophonia in individuals with PD. LSVT-BIG, on the other hand, is a protocol derived from LSVT-LOUD, used in neurorehabilitation, consisting of focused large-amplitude functional movements performed with great effort. Maximal Daily exercises consist of seven standard exercises. Functional component tasks, on the other hand, will be created for movements in which the patient has difficulty in daily life activities selected individually based on his complaints. In hierarchical tasks, daily life activities with difficulties will be studied with large amplitudes. Exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week, 60 minutes a day, 4 weeks protocol respectively.
  Arms: a) TELEREHABILITATION BASED LSVT BIG TREATMENT GROUP
Other: Telerehabilitation Based Functional Balance and Mobility Exercise — These exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week and 60 minutes a day for 4 weeks.
  Exercises will get harder with each passing week and its progression will be adjusted to the patient.
  Arms: b) TELEREHABILITATION BASED FUNCTIONAL BALANCE AND MOBILITY EXERCISES GROUP

SUMMARY:
It is planned to recruit 30 individuals with Parkinson's Disease within the scope of the study. Balance, gait, activity transfers of Parkinson's Patients will be evaluated. The study will be randomly divided into two groups. In the first group, an exercise protocol called LSVT BIG will be applied via the Zoom application with mobile phone, tablet or computer for 4 days a week for 4 weeks. This exercise protocol consists of reliable movements suitable for the conditions of patients with large amplitudes. For the other group, balance and functional mobility exercises will be applied via the Zoom application with mobile phone, tablet or computer for 4 weeks, 4 days a week. Balance, walking and activity transfer measurements will be repeated at the end of a total of 4 weeks. It is planned to include 30 patients with a diagnosis of Parkinson's Disease (PD) with a level of 1-3 according to the Hoehn-Yahr scale, who applied to the Neurology Clinic of the Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurology Training and Research Hospital. The volunteers who will participate in the study will be informed about the purpose of the study, its duration, and the possible side effects of the treatment to be applied. Primary outcome measures include Mini Best Test, Biodex balance evaluation and Kinovea for gait assessment. Dynamic balance will be evaluated with Mini-Best Test, postural stability and fall risk will be evaluated with the Biodex Balance Device. With the camera to be placed on the sagittal, 3-meter walking distances will be recorded. Colored marks will be affixed to the right and left heels. The colored marks placed will be marked on the video and the step length and walking speed will be calculated with the Kinovea motion analysis software. In the secondary evaluations, Activity Specific Balance Confidence Scale-Short Form, Sit and Stand Test Five times, Parkinson's Activity Scale, Parkinsona Specific Quality of Life Scale (PHÖ-39) will be used.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a degenerative process that affects the basal ganglia, primarily substantia nigra, and other brainstem pigmented neurons, and its main clinical symptoms are resting tremor, bradykinesia, rigidity and postural reflex disorder (1). These movement symptoms usually occur unilaterally and gradually affect the other side of the body. Gait disorders are quite common in patients with Parkinson's, and the most common disabilities during walking are reduced arm swing, step length, speed, step width, and postural control inadequacy (2). One of the characteristic movement disorders in PD is hypokinesia, in which there is a decrease in motion amplitude and speed. Hypokinesia can occur during movements such as walking, speaking, and writing. When individuals with PD try to perform or coordinate two motor tasks simultaneously, hypokinesia can occur during complex actions (3). Different exercise approaches, including musculoskeletal exercises, aerobic exercises, Nordic walking, repetitive task training, sensory cues, and balance exercises have been proposed for the treatment of movement disorders and gait in these patients (4). The LSVT BIG protocol, which consists of large-amplitude exercises for movement disorders, has been used in treatment in recent years (5). High-intensity motion amplitude training in PD was firstly implemented in the form of LSVT LOUD to improve hypophonia. The newly developed LSVT BIG treatment, derived from LSVT LOUD, aims to restore the normal range of motion by re-adjusting the patient's perception of movement and walking. Treatment focuses on intense exercise of large amplitude movements. The LSVT BIG exercise intensity was determined as 16 individualized 1-hour sessions, 4 times a week for 4 weeks. Each exercise is repeated at least 8 times and is performed with an effort of 80%, with rest breaks minimized as much as possible (6). LSVT BIG training consists of maximal daily exercises, functional component tasks, BIG walking and hierarchy tasks. The aim of the training is to readjust movement during all functional tasks in the clinic and to encourage the transfer of the newly acquired motion amplitude to all non-clinical tasks. As needed, the therapist provides visual and verbal feedback to increase the amplitude of the movement. The maximum daily exercises consist of 7 versatile standard exercises performed while sitting and standing. In the functional component tasks section, it performs 5 tasks selected according to patient goals and therapists' evaluation, these tasks are performed over and over again, focusing on increasing the amplitude of motion in each session. The BIG focuses on the patient stride length and the increasing amplitude of arm swing, and the distance is determined by walking speed and endurance. In the hierarchy tasks section, the therapist designs the functional task record form based on the patient's notification, a set of movements created based on the patient's notification, and hierarchical tasks are developed in accordance with the determined functional goals. Hierarchical tasks can be advanced by increasing the complexity of the environment. In addition, the patient is instructed to apply the acquired skills in the home environment in order to maintain the principles of this education in daily life activities (7). Although LSVT BIG treatment has been shown to have positive effects on walking speed and goal-oriented activities, its effects on freezing, balance, bed mobility and transfers during walking have not yet been specified (6). Although research on the efficacy of LSVT BIG treatment is limited, the European Physiotherapy PD Guideline recommends this exercise approach to improve walking, balance, transfers and physical capacity (8). In this guide, it is seen that exercise programs that include functional activities related to balance have an important place in the rehabilitation of PD. However, there are limited studies comparing the effectiveness of exercise types and exercise methods that can provide normal range of motion with similar intensity (9). Lack of dose-response relationships in LSVT-BIG treatment, access to the clinical environment of patients for 16 sessions and four weeks, and limitations on practical applicability of the treatment were emphasized (10). The determined standard protocol imposes a significant temporal and economic burden for outpatients (11). For this reason, it is thought that performing LSVT BIG treatment via video conferencing method and remote exercise monitoring with tele-rehabilitation, will increase the participation of patients. The implementation of remote rehabilitation interventions through telerehabilitation or communication technology is used in individuals with PD as a means of overcoming barriers and increasing compliance in many patient populations with good results. It has been shown that participation in telerehabilitation and walking exercises is higher in this population than in face-to-face exercises (12). In addition, it is stated that reduced physical exercise and increased psychological stress in the Covid 19 pandemic can worsen the symptoms of PD, and it is more important than ever to encourage home-based, adequate dose exercises. During this period, remote follow-up of individuals with PD is more reliable; It is clearly seen that online exercise, dance lessons or web-based applications for patients stand out (13). The aim of our study is to compare the effects of telerehabilitation-based LSVT-BIG protocol and telerehabilitation-based functional balance and mobility exercises in Parkinson's patients.

It is planned to include 50 patients diagnosed with Parkinson's Disease (PD) with a level of 1-3 according to the Hoehn-Yahr scale, who applied to the Neurology Clinic of Bakırköy Psychiatric and Neurological Diseases Hospital between August 2020 and September 2021. The volunteers who will participate in the study will be informed about the purpose of the study, its duration, and the possible side effects of the treatment to be applied. Their consent will be obtained with the "Informed Consent Form" prepared in accordance with the standards set by the Istanbul University Cerrahpaşa Medical Faculty Clinical Research Ethics Committee and the study will be conducted in accordance with the Declaration of Helsinki.The number of cases to be taken for each group at 80% confidence interval, considering the smallest detectable difference (Smallest Detectable Difference, SDD) 3.4, and the minimal clinical significant change (Minimal Clinically Important Difference, MCID) 3.5, among the primary outcome measures 16 was determined.

Primary outcome measures include Mini Best Test, Biodex balance evaluation and Kinovea for gait assessment. Dynamic balance will be evaluated with Mini-Best Test, postural stability and fall risk will be evaluated with the Biodex Balance Device. With the camera to be placed on the sagittal, 3-meter walking distances will be recorded. Colored marks will be affixed to the right and left heels. The colored marks placed will be marked on the video and the step length and walking speed will be calculated with the Kinovea motion analysis software. In the secondary evaluations, Activity Specific Balance Confidence Scale-Short Form, Sit and Stand Test Five times, Parkinson's Activity Scale, Parkinsona Specific Quality of Life Scale (PHÖ-39) will be used.

1. TELEREHABILITATION BASED LSVT BIG TREATMENT GROUP Lee Silverman Voice Treatment-LOUD therapy is a protocol involving intensive speech therapy, which was initiated at the Lee Silverman Parkinson Center between 1987-1989 to heal hypophonia in individuals with PD. LSVT-BIG, on the other hand, is a protocol derived from LSVT-LOUD, used in neurorehabilitation, consisting of focused large-amplitude functional movements performed with great effort. Maximal Daily exercises consist of seven standard exercises. Functional component tasks, on the other hand, will be created for movements in which the patient has difficulty in daily life activities selected individually based on his complaints. In hierarchical tasks, daily life activities with difficulties will be studied with large amplitudes (10). Exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week, 60 minutes a day, 4 weeks protocol respectively.
2. TELEREHABILITATION BASED FUNCTIONAL BALANCE AND MOBILITY EXERCISES GROUP These exercises will be applied simultaneously with the physiotherapist over the Zoom application, 4 days a week and 60 minutes a day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a definite diagnosis of Parkinson's disease according to the United Kingdom (UK) Brain Bank Criteria and being 1-3 on the Hoehn-Yahr scale
* A score of at least 21 on the Montreal cognitive assessment scale test
* To be able to walk independently on flat ground without assistive devices
* Stability of drug treatment taken in the last 1 month
* Patients are in the "on" period

Exclusion Criteria

* Serious hearing or vision problems
* Having other neurological, cardiovascular, or orthopedic impairments that can prevent walking
* Any other neurological disorder (eg dementia, cerebrovascular disease)
* Have an education level of less than 5 years
* Having vascular lower extremity pathologies
* Not having internet access with a smartphone or computer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Mini-Best Test | 15 minutes
  The Mini-BEST balance scale will be used in the assessment of dynamic balance, this scale is a one-dimensional and highly reliable measurement method with 14 items, requiring approximately 15 minutes to complete. The Mini-BEST test focuses on postural responses, dynamic gait and sensory orientation to reveal balance problems and is frequently used in Parkinson's patients. Each item is scored between 0 and 2. A score of 0 indicates that the person cannot fulfill that task, 28 points is the best indicator.
Biodex Balance Assessment | 10 minutes
  The Biodex Balance System (BBS; Biodex Medical System Inc., Shirley, NY, USA) will be used to measure the displacement of the center of foot pressure (CoP). Biodex Balance System 20 Hz. It consists of a circular platform that allows 20 degrees of platform tilt in a range of 360 degrees of motion at sampling rate. Measures of postural stability score for BBS; It is in the form of the General Stability Index (OSI), Medial-Lateral Stability Index (MLSI) and Anterior-Posterior Stability Index (APSI). The degree of unbalance of the surface can be adjusted from the most stable (level 8) to the least stable levels (level 1)
Kinovea Gait Analysis | 15 minutes
  3 meters walking distance will be recorded with the camera to be placed in the sagittal. Colored markings will be affixed to the right and left heels. The colored marks placed will be marked on the video and step lengths, walking speed and arm swing will be calculated with the Kinovea motion analysis software. The video will express the cadence (number of steps per minute), right and left stride lengths
Timed Up and Go (TUG) Test | 10 minutes
  Timed Up and Go (TUG) test is a simple, widely used and rapid test to evaluate mobility, balance and fall risk. To perform the test, participants must stand up from a standard chair, walk comfortably 3 meters from the ground, turn and return to the chair, and sit on the same chair. All steps of the test will be measured using a stopwatch

SECONDARY OUTCOMES:
Activity Specific Balance Confidence Scale - Short Form: | 5 minutes
  The short form of Activity Specific Balance Confidence Scale will be used to measure patients' balance confidence. Activity-Specific Balance Confidence Scale is answered with the self-perception of the individual, which consists of 16 items. It includes values in the range of 0-100 and measures the perceived ability to maintain balance under different conditions. The highest score indicates full confidence in their balance abilities. The short form of this scale consists of 6 questions of the original version of the scale and it has been stated that it is valid and reliable when associated with the risk of falling in the PD population.
Five Times Sit & Stand Test | 5 minutes
  This test will be used in our study to determine repetitive motion performance. Individuals will be instructed to cross their arms over their chest and sit down to rest their back against the back of the chair. He will be asked to sit and stand five times as soon as possible, and then time will be recorded. The performance of this test in individuals with PD has been found to be associated with balance and bradykinesia and has been recommended as a reliable method
Parkinson Activity Scale | 15 minutes
  It is a scale developed to evaluate the functional status in PD. It consists of a total of 10 items, including the sections of standing up from the chair, walking akinesia and in-bed mobilization, and provides information about the transfer status of the patients. Evaluations are made between 0 and 4, and a high score is an indicator of good performance
Parkinson-Specific Quality of Life Scale | 15 minutes
  The Parkinson-Specific Quality of Life Scale will be used in quality of life assessment. PDQ-39 is a self-report questionnaire that uses the 5-point Likert scale to assess the quality of life such as the severity of symptoms of mobility, daily living activities, emotional well-being, social support, cognition, and communication. The total score is between 0-100, and the higher the score indicates that the quality of life is at a lower level

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersoz Huseyinsinoglu, Assoc.Prof, Study Director — Istanbul University - Cerrahpasa; Nazan Karagoz Sakallı, MD, Study Chair — Bakırköy Prof.Dr. Mazhar Osman Psychiatric and Neurological Diseases Hospital; Aysu Sen, Assoc.Prof., Study Chair — Bakırköy Prof.Dr. Mazhar Osman Psychiatric and Neurological Diseases Hospital
Locations (1):
- Bakırköy Prof.Dr. Mazhar Osman Psychiatric and Neurological Diseases Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebersbach G, Grust U, Ebersbach A, Wegner B, Gandor F, Kuhn AA. Amplitude-oriented exercise in Parkinson's disease: a randomized study comparing LSVT-BIG and a short training protocol. J Neural Transm (Vienna). 2015 Feb;122(2):253-6. doi: 10.1007/s00702-014-1245-8. Epub 2014 May 29. PMID 24872078
- [Background] Millage B, Vesey E, Finkelstein M, Anheluk M. Effect on Gait Speed, Balance, Motor Symptom Rating, and Quality of Life in Those with Stage I Parkinson's Disease Utilizing LSVT BIG(R). Rehabil Res Pract. 2017;2017:9871070. doi: 10.1155/2017/9871070. Epub 2017 Feb 26. PMID 28331638
- [Background] Strouwen C, Molenaar EALM, Munks L, Keus SHJ, Zijlmans JCM, Vandenberghe W, Bloem BR, Nieuwboer A. Training dual tasks together or apart in Parkinson's disease: Results from the DUALITY trial. Mov Disord. 2017 Aug;32(8):1201-1210. doi: 10.1002/mds.27014. Epub 2017 Apr 25. PMID 28440888
- [Background] Strouwen C, Molenaar EA, Keus SH, Munks L, Munneke M, Vandenberghe W, Bloem BR, Nieuwboer A. Protocol for a randomized comparison of integrated versus consecutive dual task practice in Parkinson's disease: the DUALITY trial. BMC Neurol. 2014 Mar 27;14:61. doi: 10.1186/1471-2377-14-61. PMID 24674594
- [Background] van der Kolk NM, King LA. Effects of exercise on mobility in people with Parkinson's disease. Mov Disord. 2013 Sep 15;28(11):1587-96. doi: 10.1002/mds.25658. PMID 24132847
- [Background] Janssens J, Malfroid K, Nyffeler T, Bohlhalter S, Vanbellingen T. Application of LSVT BIG intervention to address gait, balance, bed mobility, and dexterity in people with Parkinson disease: a case series. Phys Ther. 2014 Jul;94(7):1014-23. doi: 10.2522/ptj.20130232. Epub 2014 Feb 20. PMID 24557655
- [Background] Fishel SC, Hotchkiss ME, Brown SA. The impact of LSVT BIG therapy on postural control for individuals with Parkinson disease: A case series. Physiother Theory Pract. 2020 Jul;36(7):834-843. doi: 10.1080/09593985.2018.1508260. Epub 2018 Aug 17. PMID 30118624
- [Background] Domingos J, Keus SHJ, Dean J, de Vries NM, Ferreira JJ, Bloem BR. The European Physiotherapy Guideline for Parkinson's Disease: Implications for Neurologists. J Parkinsons Dis. 2018;8(4):499-502. doi: 10.3233/JPD-181383. PMID 30149464
- [Background] Fox C, Ebersbach G, Ramig L, Sapir S. LSVT LOUD and LSVT BIG: Behavioral Treatment Programs for Speech and Body Movement in Parkinson Disease. Parkinsons Dis. 2012;2012:391946. doi: 10.1155/2012/391946. Epub 2012 Mar 15. PMID 22530161
- [Background] Ellis T, Latham NK, DeAngelis TR, Thomas CA, Saint-Hilaire M, Bickmore TW. Feasibility of a virtual exercise coach to promote walking in community-dwelling persons with Parkinson disease. Am J Phys Med Rehabil. 2013 Jun;92(6):472-81; quiz 482-5. doi: 10.1097/PHM.0b013e31828cd466. PMID 23552335
- [Background] Helmich RC, Bloem BR. The Impact of the COVID-19 Pandemic on Parkinson's Disease: Hidden Sorrows and Emerging Opportunities. J Parkinsons Dis. 2020;10(2):351-354. doi: 10.3233/JPD-202038. No abstract available. PMID 32250324
- [Result] McDonnell MN, Rischbieth B, Schammer TT, Seaforth C, Shaw AJ, Phillips AC. Lee Silverman Voice Treatment (LSVT)-BIG to improve motor function in people with Parkinson's disease: a systematic review and meta-analysis. Clin Rehabil. 2018 May;32(5):607-618. doi: 10.1177/0269215517734385. Epub 2017 Oct 5. PMID 28980476
- [Derived] Kaya Aytutuldu G, Ersoz Huseyinsinoglu B, Karagoz Sakalli N, Sen A, Yeldan I. LSVT(R) BIG versus progressive structured mobility training through synchronous telerehabilitation in Parkinson's disease: A randomized controlled trial. Neurol Sci. 2024 Jul;45(7):3163-3172. doi: 10.1007/s10072-024-07322-0. Epub 2024 Jan 25. PMID 38267603